CLINICAL TRIAL: NCT00235937
Title: An Open, Phase II Trial Assessing the Objective Response Rate After Combination of Arimidex® 1mg Per os/Day and Zoladex® 3.6 mg Sub Cut/Monthly as 1st Treatment for Premenopausal Receptor Positive Advanced or Metastatic Breast Cancer
Brief Title: Study on Pre-menopausal Patients With Advanced ER and PR + BC Treated With Arimidex Plus Zoladex
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5390L00061 Roche Study; THR 0104233 C
Record Dates: First submitted 2005-10-10; First posted 2005-10-12 (Estimated); Last update posted 2011-01-21 (Estimated); Status verified 2011-01

CONDITIONS: Breast Cancer
Keywords: Premenopausal; Advanced Breast Cancer; Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Goserelin

INTERVENTIONS:
Drug: Anastrozole and goserelin

SUMMARY:
The purpose of this study is to determine the efficacy and tolerance of the association of two drugs already marketed and used to treat your disease: Arimidex® 1 Mg per day per os and Zoladex® 3,6 Mg in injections under cutaneous once per month in subjects with breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent, premenopausal women 18 years or older, histologically or cytologically confirmed locally advanced or metastatic breast cancer, suitable for endocrine treatment, no curative treatment available,, one or more measurable lesions, life expectancy more than 6 months, normal biological parameters.

Exclusion Criteria:

* Presence of life-threatening metastases, previous endocrine therapy or chemotherapy for advanced or metastatic disease, any previous treatment with hormone (LH-RH) severe or uncontrolled systemic disease, pituitary adenoma, High risk of medullar compression.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2001-12; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility and efficacy of the combination of these 2 drugs in these patients

SECONDARY OUTCOMES:
To assess clinical benefit rate, time to progression, duartion of response and safety in patients treated with the combination of these 2 drugs

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (7):
- France (7):
  - Angers
  - Caen
  - Poitiers
  - Rennes
  - Rouen
  - Saint-Herblain
  - Toulouse